CLINICAL TRIAL: NCT00560014
Title: Role of Immunonutrient Levels in Preventing Complications After Renal Transplantation
Brief Title: Nutrient Levels Alter Transplant Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: LIPIDS; R03 AI142743; 5U01AI040167 (NIH)
Record Dates: First submitted 2007-11-14; First posted 2007-11-19 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Arginine; Rapeseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Arginine and Canola oil supplemented group
  Interventions: Dietary Supplement: Arginine and canola oil
- 2 (Experimental): Arginine and Coromega
  Interventions: Dietary Supplement: Coromega and Arginine
- 3 (No Intervention): Control

INTERVENTIONS:
Dietary Supplement: Arginine and canola oil — Canola oil 1 tablespoon BID Arginine 9.0grams BID
  Other Names: Arginaid
  Arms: 1
Dietary Supplement: Coromega and Arginine — Arginine 9.0 grams BID Coromega dose based on weight
  Other Names: Arginaide
  Arms: 2

SUMMARY:
The purpose of this study is to look at lipid profiles of plasma and RBC and amino acid profiles in plasma to determine if they are associated with allograft rejection, calcineurin inhibitor toxicity or new onset diabetes mellitus in renal transplant patients receiving dietary supplements with arginine and omega-3 fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipient
* Appropriate blood samples drawn and analyzed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1997-09; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Plasma and red blood cell lipid profiles | Within 1 year
Plasma amino acid profiles | within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: J. W. Alexander, M.D., Principal Investigator — UC Surgeons Center fo Surgical Weight Loss/ University of Cincinnati
Locations (2):
- United States (2):
  - Washington Hospital, Washington D.C., District of Columbia
  - Duke University School Of Medicine, Durham, North Carolina

REFERENCES:
- [Derived] Alexander JW, Goodman HR, Succop P, Light JA, Kuo PC, Moser AB, James JH, Woodle ES. Influence of long chain polyunsaturated fatty acids and ornithine concentrations on complications after renal transplant. Exp Clin Transplant. 2008 Jun;6(2):118-26. PMID 18816238